CLINICAL TRIAL: NCT05986279
Title: Improving Psychological and Vestibular Health Using a Novel Intervention: The Making Informed Decisions in Gaze and Postural Stability (MINDGAPS) System
Brief Title: Improving Psychological and Vestibular Health: MINDGAPS
Acronym: MINDGAPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Montana (Other)
Collaborators: United States Naval Medical Center, San Diego (U.S. Federal Agency); Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Brian Loyd, Professor, University of Montana
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 168-22
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Vestibular Hypofunction
Keywords: Rehabilitation; mild traumatic brain injury; dynamic visual acuity; gaze stability; postural stability; dizziness; psychological health
MeSH Terms: conditions — Brain Concussion; Dizziness; Psychological Well-Being | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: One group is enrolled into a longitudinal, single group intervention using vestibular rehab. The other group is enrolled as a cross-sectional observational assessment used for developing normative data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehab (Experimental): 6 weeks of vestibular physical therapy guided by the use of the MINDGAPS decision support system
  Interventions: Other: Rehab
- Observational (No Intervention): Normative data development of performance on vestibular measures following mTBI

INTERVENTIONS:
Other: Rehab — 6 weeks of vestibular rehabilitation guided by the MINDGAPS decision support system
  Arms: Rehab

SUMMARY:
The purpose of this study is twofold: 1) Develop norms for measures of inner ear function and psychological health, and 2) Examine the feasibility of using the MINDGAPS system (a remote monitoring system) to track progress during physical therapy or rehabilitation for inner ear problems following a concussion or mild Traumatic Brain Injury.

DETAILED DESCRIPTION:
The intersection between vestibular disturbance and psychological health provides a unique clinical opportunity to address both the modifiable symptoms of vestibular disturbance as well as psychological health. This project aims to advance our understanding of the causal link between vestibular disturbance and poor psychological health and aligns directly with the Traumatic Brain Injury and Psychological Health Research Program (Funding Opportunity: W81XWH-21-TBIPHRP-TRA). Specifically, the proposed research is responsive to each of the three focus areas: Understand- this project is designed to advance the understanding of an established link between vestibular disturbance (e.g., dizziness and poor balance) and poor psychological health (e.g., anxiety, depression, and social isolation) in survivors of mild traumatic brain injury (mTBI). Prevent- the MINDGAPS system allows for precise assessment of dynamic visual acuity (computerized dynamic visual acuity [cDVA]) and postural sway (instrumented balance accelerometry measure [iBAM]), two objective and extensively validated surrogates of vestibular health. Additionally, MINDGAPS uses these measures to inform care decisions via a user-friendly web application. Treat- vestibular assessment is key to effective vestibular care, as it allows for personalization of treatment programs and monitoring progress over time.

Objective/Hypothesis:

The overall objective of this project is two-fold: 1) Test the preliminary efficacy of the MINDGAPS system to improve psychological health and vestibular disturbance in active-duty and Veteran Service Members (SM) with history of mTBI and 2) refine the MINDGAPS system by developing military-specific normative data and using Community-Based Participatory Research (CBPR) to incorporate the lived experiences of mTBI survivors, their caregivers, and clinicians in the design of the MINDGAPS technology and intervention.

Specific Aims:

Specific Aim 1 (Preliminary Efficacy): Examine the preliminary efficacy of the MINDGAPS system to improve psychological and vestibular health in active-duty and Veteran SM with sub-acute and chronic mTBI.

Specific Aim 2 (Military-specific Normative Data): Collect a cross-sectional sample of cDVA, iBAM, and other relevant measures in active-duty and Veteran Service Members across three different stages of mTBI-no diagnosed history of mTBI, sub-acute mTBI (2-6 months), and chronic mTBI (>6 months)-for the development of normative values in military-specific populations.

Specific Aim 3 (Refinement of MINDGAPS): Utilize CBPR to refine and improve the MINDGAPS system for different stakeholders (SM, caregivers, and clinicians) and position MINDGAPS for examination in a large-scale clinical trial as well as translation into clinical practice.

Study Design:

Aim 1: Using a single-cohort (N=36) double-baseline design, all participants will be tested twice during a no-intervention baseline period, then once following a 6-week course of vestibular training with the MINDGAPS system. Efficacy will be determined by comparing change during the baseline period to change over the course of the intervention period. Aim 2: A large sample of active-duty and Veteran SM (N=300) will be tested in a single, cross-sectional assessment to build military-specific normative vestibular data. Aim 3: We will use a convergent mixed-methods analysis of study participant feedback, in combination with quantitative results and stakeholder engagement, to drive refinement of the MINDGAPS system throughout the study period.

Impact:

Signs of vestibular disturbance are the most commonly reported symptoms following mTBI, and vestibular disturbance is causally implicated in the development of poor psychological health following mTBI. Interventions aimed at improving vestibular disturbance can improve debilitating symptoms such as poor balance and dizziness. The completion of this study will move MINDGAPS to a technology readiness level of 8, preparing it to be studied in a large clinical trial in the next phase of work.

Relevance to Military Health:

Interventions aimed at improving vestibular disturbance would have profound impacts on both active-duty SM (inability to visually focus during dynamic tasks- e.g., field of fire) and Veterans (increased risk of falls). Furthermore, the MINDGAPS system enables rapid and precise assessment of vestibular functioning at low cost and therefore has tremendous potential to enhance the delivery of clinical services within a number of active-duty environments including far-forward military settings or Veterans living in rural areas.

ELIGIBILITY:
Inclusion Criteria:

* Veteran or Active Duty Military Service Member
* Ability to stand independently
* Legally autonomous and able to self-consent

Exclusion Criteria:

* Acute head injury (within the previous 2 months)
* History of moderate or severe head injury (i.e., loss of consciousness greater than 30 minutes or post-traumatic amnesia greater than 1 day)
* Current diagnosis of spine disorders in the neck
* Diagnosis of problems with the arteries in your neck
* Blindness
* If you have been diagnosed with abnormal eye movements (also called "ocular motor palsy")
* If you have previously had a stroke or been diagnosed with a neurodegenerative disorder ( e.g., Parkinson's Disease, Multiple Sclerosis)
* If you have been previously diagnosed primary vestibular dysfunction ( e.g., congenital peripheral vestibular syndrome)
* If you have previously been diagnosed with a brain tumor
* If you are currently receiving physical therapy care for balance or dizziness problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2027-09-29 (Estimated); Study Completion 2027-09-29 (Estimated)

PRIMARY OUTCOMES:
Computerized Dynamic Visual Acuity (cDVA) | through study completion, an average of 12 weeks
  computerized measure of functional gaze stability

SECONDARY OUTCOMES:
Instrumented postural sway assessment | through study completion, an average of 12 weeks
  instrumented assessment of static postural stability
Video head impulse testing (vHIT) | through study completion, an average of 12 weeks
  computerized assessment of vestibulo-ocular reflex function
Functional Gait Assessment (FGA) | through study completion, an average of 12 weeks
  The Functional Gait Assessment (FGA) is a 10-item measure that examines dynamic stability during various walking tasks on a marked 6-m (20-ft) length and 12-inch wide walkway. Each item is rated from 0-3 with higher scores indicating better dynamic stability. Tasks within the FGA require head and/or body motion during walking activities which will be assessed using body-worn 3D inertial measurement units
Dizziness Handicap Inventory (DHI) | through study completion, an average of 12 weeks
  The DHI is a self assessment inventory designed to evaluate the self-perceived handicap effects imposed by dizziness or unsteadiness and has documented test-retest and internal consistency reliability. The DHI consists of 25 questions subgroup into functional, emotional, and physical components. The total score ranges from 0-100, with higher scores indicating greater handicap.
Life Space Mobility Assessment (LSA) | through study completion, an average of 12 weeks
  patient reported questionnaire examining community mobility. The maximum possible score is 40 with higher scores indicating better life space mobility.
Role Participation Questionnaire | through study completion, an average of 12 weeks
  patient reported questionnaire assessing participant role in society. The questionnaire asks 17 questions with lower scores indicating greater societal role.
General Well Being Scale | through study completion, an average of 12 weeks
  patient reported questionnaire assessing psychological health. Consists of 18 questions with scores ranging from 0-110 and higher scores indicating better well-being.
Healthcare Utilization Questionnaire | through study completion, an average of 12 weeks
  patient reported questionnaire assessing participants use of healthcare.
Self-Administered Comorbidity Questionnaire (SCQ) | through study completion, an average of 12 weeks
  patient reported questionnaire assessing health related problems, treatment and limitations.
Military Service Information (MSI) | through study completion, an average of 12 weeks
  patient reported questionnaire inquiring about military service
Ohio State University Head Injury History | through study completion, an average of 12 weeks
  patient reported questionnaire assessing injuries to head and neck
Primary Care 5-Item PTSD Screen | through study completion, an average of 12 weeks
  patient reported questionnaire to identify individuals with probable PTSD
Visual Analogy Scale of Dizziness and Unsteadiness | through study completion, an average of 12 weeks
  patient report of severity of dizziness and unsteadiness. Participants are asked to draw a single line on a 10 cm line with a higher number indicating greater dizziness or unsteadiness.
High-Level Mobility Assessment (HiMT) | through study completion, an average of 12 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Naval Medical Center San Diego, San Diego, California
  - University of Montana, Missoula, Montana